CLINICAL TRIAL: NCT01547923
Title: The Medical-financial Evaluation of Pre-therapeutic Screening by a Joint Phenotypic-pharmacogenetic Approach for Metabolic Fluoropyrimidine Enzyme Deficiency in Terms of Serious Toxicity Risk Prevention : a Multicentric Case Study
Brief Title: Pre-therapeutic Identification of Dihydropyrimidine Dehydrogenase Gene (DPD) Deficiency for Predicting Toxicity to Fluoropyrimidines
Acronym: DPD côlon
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study stopped due to a death in the arm control
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CPP-380; 2008-000026-39 (EudraCT Number)
Record Dates: First submitted 2012-02-28; First posted 2012-03-08 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Colorectal Cancer; Intravenous 5 Fluorouracile
Keywords: Colorectal Cancer; DihydroPyrimidine Dehydrogenase; Lethal toxicity; Fluoropyrimidine
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A : pre-therapeutic screening for DPD deficiency (Experimental): Prior to treatment by fluoropyrimidines,a DPD deficiency is identified by a joint phenotypic-pharmacogenetic approach.
  Interventions: Genetic: Blood sample for phenotypic and pharmacogenetic analysis.
- B : no pretherapeutic research of DPD deficiency (Other): For patients included in this arm, a blood sample will be taken prior to treatment by fluoropyrimidines but not analysed. If grade 3 or 4 toxicity levels are encountered during treatment, DPD deficiency will be detected.
  Interventions: Genetic: Blood sample for phenotypic and pharmacogenetic analysis.

INTERVENTIONS:
Genetic: Blood sample for phenotypic and pharmacogenetic analysis. — Prior to treatment by 5-FU, a DPD deficiency is identified thanks to just one blood sample (lithium heparinate).
  Arms: A : pre-therapeutic screening for DPD deficiency
Genetic: Blood sample for phenotypic and pharmacogenetic analysis. — Blood sample (lithium heparinate) will be taken prior to treatment but not analysed.
  Arms: B : no pretherapeutic research of DPD deficiency

SUMMARY:
The aim of this study is to demonstrate the medical and financial benefit of pre-therapeutic screening of DPD deficiency for predicting toxicity to fluoropyrimidines.

DETAILED DESCRIPTION:
The fluoropyrimidines, of which 5-Fluorouracil is the most important, represent a family of medication that is used in particular in cancerology. They are molecules widely used in cancerology since they can be found in nearly 45% of chemotherapy protocols and in the treatment of about 50% of cancers (colorectum, oesophagus, stomach, breast, upper digestive and respiratory tracts). They are not only used in metastatic situations but also more and more in adjuvant situations, in other words for patients treated for a localised tumour, presenting a risk of relapse. A severe toxic risk cannot be tolerated in these conditions, and the doctor should assure the maximum level of safety for his patients. These medicines are the cause of 3% of grade IV toxicity from the first or second administration, and for 0.3% of deaths. To this one can add on a total of 20 to 25% grade III-IV toxic events.

Anticancer treatment is mostly administered by body size and in the best of cases after a few basic biological examinations such as a haemogram and renal status, without taking into consideration any individual particularities, whether genetic or epigenetic. Among potential toxicity risk factors one can find individual metabolic differences linked to genetic modifications of metabolism enzymes as well as differences in the chemical receptors and transporters.

For fluoropyrimidines, a polymorphism was found for the dihydropyrimidine dehydrogenase gene (DPD), a major catabolism enzyme. A deficit of this enzyme is a major counter-indication for the use of these medicines.

Early determination of DPD status would allow identification of patients at risk and would thus help in subsequent dose adjustment or selection of other treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer, histologically confirmed, with all types included (including adjuvant cases), requiring treatment with intravenous 5-fluorouracil.
* anterior chemotherapy authorised, with the exception of chemotherapy containing a derivate of 5-Fluorouracil
* Age > or = 18 years
* WHO Performance status < or = 2
* Haematologic and hepatic parameters : neutrophils > or = 1000 /mm3, platelets > or = 100000/mm3, Total bilirubin < or = 2 x ULN, AST and ALT < or = 3 x ULN, APL < or = 5 x ULN
* Complete initial assessment before first treatment administration for imaging and pharmacogenetic, within 15 days for biology, and within 7 days for clinical examination.
* Signed written informed consent

Exclusion Criteria:

* Prior chemotherapy with fluoropyrimidines
* Symptomatic or uncontrolled ventral nervous system metastases
* Psychiatric Disease disrupting the trial understanding and the enlightened and voluntary consent character
* Patient who is pregnant or breast feeding
* Woman not consenting to use adequate contraceptive precautions during the study
* Patient who can not submit itself to the formal follow-up for psychological, social, family or geographical reasons
* Significant serious pathology or any instable medical condition (cardiac pathology uncontrolled, myocardial infarction within 6 months before enrollment, systemic active uncontrolled infection)
* any investigational agent within 4 weeks before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1142 (Actual)
Dates: Start 2008-06-16 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03-04 (Actual)

PRIMARY OUTCOMES:
Number and nature of grade IV toxicity. | Up to 4 weeks.
  The percentage of severe toxicity (grade IV) will be analyzed in each arm. We expect a reduction of the early, severe, grade IV acute side-effects from 3% to 0.6% in the detected group with adapted doses.

SECONDARY OUTCOMES:
Number of grade III-IV toxic events. | Up to 6 months.
  We expect a reduction of the number of grade III-IV toxic events, whenever they occur, from 25% to 5% in the detected group with adapted doses.
Mortality rate. | up to 6 months.
  The current mortality rate of 3 per thousand patients will be cut to 0 in the detected group with adapted doses.
Medical-financial study of pre-therapeutic screening. | Up to 6 months.
  We will carry out a comparison of the prevention costs and the costs related to treating patients with toxicity. Direct costs and indirect costs will be taken into account.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Capitain, MD, PhD, Principal Investigator — Institut Cancerologie de l'Ouest
Locations (25):
- France (25):
  - ICO Paul Papin, Angers
  - CHU Jean Minjoz, Besançon
  - CHU Morvan, Brest
  - CHU Côte de Nacre, Caen
  - Centre François Baclesse, Caen
  - Pôle Santé Léonard de Vinci, Chambray-lès-Tours
  - Centre Hospitalier du Haut Anjou, Château-Gontier
  - Centre Hospitalier, Cholet
  - Clinique des Cèdres, Cornebarrieu
  - Hôpital Henri Mondor, Créteil
  - CH Sarthe et Loir, La Flèche
  - Centre Hospitalier Les oudairies, La Roche-sur-Yon
  - Centre Hospitalier, Laval
  - Centre Hospitalier, Le Mans
  - Centre Oscar Lambret, Lille
  - Centre d'oncologie de Gentilly, Nancy
  - CHU Hotel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - HEGP, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - ICO René Gauducheau, Saint-Herblain
  - Centre Hospitalier, Saumur
  - Institut Claudius Regaud, Toulouse
  - Hôpital Purpan, Toulouse
  - CHU Trousseau, Tours